CLINICAL TRIAL: NCT03442738
Title: A Prospective Randomized Comparison of the Adenoma Detection Rate in Screening Colonoscopy With and Without a Disposable Cap (ENDOCUFF VISION®)
Brief Title: A Prospective Randomized Comparison of the Adenoma Detection Rate With a Disposable Cap (ENDOCUFF VISION®)
Acronym: Endocuff
Status: Completed | Type: Observational
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Collaborators: Norgine (Industry)
Responsible Party: Principal Investigator, Prof. Dr. Thomas Rösch, Prof. Dr. med., Universitätsklinikum Hamburg-Eppendorf
Other Study IDs: PV 5294
Record Dates: First submitted 2018-02-02; First posted 2018-02-22 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Adenoma Detection Rate
Keywords: ADR; adenoma; polyp; colon; screening; colorectal carcinoma (CRC); cap; endoscopy; colonoscopy; private practice
MeSH Terms: conditions — Adenoma; Polyps; Colorectal Neoplasms; Anterior polar cataract 2

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group I Endocuff group: Group I Endocuff cap use
  Interventions: Procedure: Endocuff group
- Group II standard colonoscope: Group II standard colonoscope, no further device used
  Interventions: Procedure: Endocuff group

INTERVENTIONS:
Procedure: Endocuff group — Endocuff Vision cap on Standard colonoscope

SUMMARY:
The aim of this study is to evaluate the effect of ENDOCUFF VISION® (caps with soft, about 1 cm long lateral feet of rubber ("Endocuff") to flatten the colon folds) on ADR in a real-life setting (general practices) and in a homogenous patient collective (screening colonoscopies only).

It is a prospective randomized multi centric study, with participation of at least 10 study sites (private practice). The study is an inverstigator-initiated trial (IIT).

Depending on the randomization (closed envelope), the patients are examined with the standard instruments without or with ENDOCUFF VISION®.

Group 1: screening colonoscopy with standard colonoscopes with ENDOCUFF VISION® Group 2: screening colonoscopy with standard colonoscopes without cap

DETAILED DESCRIPTION:
Colonoscopy is currently the best method for the detection of colon carcinomas and, as precursor, adenomas, since these can also be biopsied and removed. Therefore, the screening colonoscopy was introduced at the end of 2002 (covered by state insurance) from the age of 55. The main quality parameter for outcome quality is the adenoma detection rate (ADR), which correlates with the rate of the carcinomas prevented. However, since even smaller polyps, especially if they are flat or sunken, may be relevant for colon cancer development, the aim of colonoscopy should be to be able to recognize and remove as many adenomas as possible. There is a need to optimize the efficiency of screening colonoscopy by increasing the rate of adenoma detection, as it is known from many studies that approximately 15-30% of adenomas can be missed- even though the adenoma rate in the German screening colonoscopy register continues to increase over the years and currently stands at 28%.

Previous studies on the increase of the adenoma detection rate by endoscopy concerning newer endoscope technologies including conventional caps have been almost entirely negative.

For about 2 years, a newer version of ENDOCUFF VISION® caps (caps with soft, about 1 cm long lateral feet of rubber (Endocuff) to flatten the colon folds) is available which has already been used in about 8,000 colonoscopies in Germany and another 10,000 colonoscopies in Europe; there are no studies on this version of Endocuff caps.

The aim of this study is to evaluate the effect of ENDOCUFF VISION® in a real-life setting (general practices) and in a homogenous patient collective (screening colonoscopies only).

It is a prospective randomized multi centric study, with participation of at least 10 study sites (private practice). The study is an inverstigator-initiated trial (IIT).

A new technique for ADR improvement within colonoscopy can only be tested in a comparative study in two groups comparing the adenoma rate between the two groups. An independent gold standard does not exist in this sense, but the confirmation by the endoscopically taken histology serves as gold standard for the diagnosis adenoma. The alternative of double examinations (tandem colonoscopy) in each patient is in the setting of private practice not feasible.

Depending on the randomization (closed envelope), the patients are examined with the standard instruments without or with ENDOCUFF VISION®.

Group 1: screening colonoscopy with standard colonoscopes with ENDOCUFF VISION® Group 2: screening colonoscopy with standard colonoscopes without cap

ELIGIBILITY:
Inclusion Criteria:

* > 55 years
* who voluntarily undergo a screening colonoscopy
* information and signed declaration of consent

Exclusion Criteria:

* symptoms that may indicate a colonic disease
* rectal/colonic bleeding
* known colon disease for further diagnosis, e.g. Carcinoma, polyps for erosion, inflammatory bowel disease, stenosis
* follow-up/surveillance after colon carcinoma surgery or polypectomy
* anticoagulant drugs that make a biopsy or polypectomy impossible
* poor general condition (from ASA (American Society of Anesthesiologists Classification) III)
* partial/incomplete colonoscopy planned

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Screening Population for Adenoma and CRC
Sampling Method: Non-Probability Sample
Enrollment: 1382 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Adenoma Detection Rate (ADR) in the two study groups | through study completion, an average of 1 year
  Differences in ADR with or without the new disposable ENDOCUFF VISION® cap. Hypothesis: Endocuff Vision improves the adenoma detection rate (ADR) by about 25% compared to the comparison group.

SECONDARY OUTCOMES:
ADR (all adenoma/all patients) | 12 months
  ADR (all adenoma/all patients)
assessment of adenoma subgroups by location | 12 months
  differences in adenoma subgroups (between intestinal folds with good accessibility, between intestinal folds with poor accessibility, on top of intestinal fold, behind intestinal fold )
assessment of adenoma subgroups by size | 12 months
  measured by comparison with size of snare or forceps
assessment of adenoma subgroups by form | 12 months
  stem-based, broad-based, flat adenoma
assessment of adenoma subgroups by histology | 12 months
  loiw grade intraepithelial neoplasia (LGIN), high grade intraepithelial neoplasia (HGIN), sessile serrated Adenoma (SSA), Carcinoma
assessment of adenoma subgroups by adjustability | 12 months
  adjustability of adenoma by colonoscope on a score scale from 1(very good) - 6 (poor)
assessment of adenoma subgroups by resection practice | 12 months
  resection of adenoma by biopsy, polypectomy, resection by forceps, none
Intervention times | through study completion, an average of 1 year
  duration of Intervention
procedure technique | through study completion, an average of 1 year
  technical aspects of polypectomy/biopsy

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Rösch, Principal Investigator — Universitätsklinikum Hamburg-Eppendorf
Locations (9):
- Germany (9):
  - Gastroenterologische Spezialpraxis am Wittenbergplatz, Berlin
  - Gemeinschaftspraxis Hohenzollerndamm, Berlin
  - Gastroenterologie am Bayerischen Platz, Berlin
  - Praxis Dr. Mayr, Berlin
  - Praxis für Gastroenterologie in Berlin Reinickendorf, Berlin
  - Praxis Dr. med. Jens Aschenbeck, Berlin
  - Gastropraxis Eppendorfer Baum, Hamburg
  - Schwerpunktpraxis CCB Bergedorf, Hamburg
  - Magen-Darm-Zentrum, Facharztzentrum Eppendorf, Hamburg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kaminski MF, Regula J, Kraszewska E, Polkowski M, Wojciechowska U, Didkowska J, Zwierko M, Rupinski M, Nowacki MP, Butruk E. Quality indicators for colonoscopy and the risk of interval cancer. N Engl J Med. 2010 May 13;362(19):1795-803. doi: 10.1056/NEJMoa0907667. PMID 20463339
- [Background] Corley DA, Jensen CD, Marks AR, Zhao WK, Lee JK, Doubeni CA, Zauber AG, de Boer J, Fireman BH, Schottinger JE, Quinn VP, Ghai NR, Levin TR, Quesenberry CP. Adenoma detection rate and risk of colorectal cancer and death. N Engl J Med. 2014 Apr 3;370(14):1298-306. doi: 10.1056/NEJMoa1309086. PMID 24693890
- [Background] Bretagne JF, Ponchon T. Do we need to embrace adenoma detection rate as the main quality control parameter during colonoscopy? Endoscopy. 2008 Jun;40(6):523-8. doi: 10.1055/s-2007-995786. Epub 2008 May 8. No abstract available. PMID 18464196
- [Background] van Rijn JC, Reitsma JB, Stoker J, Bossuyt PM, van Deventer SJ, Dekker E. Polyp miss rate determined by tandem colonoscopy: a systematic review. Am J Gastroenterol. 2006 Feb;101(2):343-50. doi: 10.1111/j.1572-0241.2006.00390.x. PMID 16454841
- [Background] Brenner H, Altenhofen L, Kretschmann J, Rosch T, Pox C, Stock C, Hoffmeister M. Trends in Adenoma Detection Rates During the First 10 Years of the German Screening Colonoscopy Program. Gastroenterology. 2015 Aug;149(2):356-66.e1. doi: 10.1053/j.gastro.2015.04.012. Epub 2015 Apr 22. PMID 25911510
- [Background] Moriyama T, Uraoka T, Esaki M, Matsumoto T. Advanced technology for the improvement of adenoma and polyp detection during colonoscopy. Dig Endosc. 2015 Apr;27 Suppl 1:40-4. doi: 10.1111/den.12428. PMID 25556542
- [Background] Omata F, Ohde S, Deshpande GA, Kobayashi D, Masuda K, Fukui T. Image-enhanced, chromo, and cap-assisted colonoscopy for improving adenoma/neoplasia detection rate: a systematic review and meta-analysis. Scand J Gastroenterol. 2014 Feb;49(2):222-37. doi: 10.3109/00365521.2013.863964. Epub 2013 Dec 16. PMID 24328858
- [Background] Nagorni A, Bjelakovic G, Petrovic B. Narrow band imaging versus conventional white light colonoscopy for the detection of colorectal polyps. Cochrane Database Syst Rev. 2012 Jan 18;1(1):CD008361. doi: 10.1002/14651858.CD008361.pub2. PMID 22258983
- [Background] Biecker E, Floer M, Heinecke A, Strobel P, Bohme R, Schepke M, Meister T. Novel endocuff-assisted colonoscopy significantly increases the polyp detection rate: a randomized controlled trial. J Clin Gastroenterol. 2015 May-Jun;49(5):413-8. doi: 10.1097/MCG.0000000000000166. PMID 24921209
- [Background] Floer M, Biecker E, Fitzlaff R, Roming H, Ameis D, Heinecke A, Kunsch S, Ellenrieder V, Strobel P, Schepke M, Meister T. Higher adenoma detection rates with endocuff-assisted colonoscopy - a randomized controlled multicenter trial. PLoS One. 2014 Dec 3;9(12):e114267. doi: 10.1371/journal.pone.0114267. eCollection 2014. PMID 25470133
- [Background] van Doorn SC, van der Vlugt M, Depla A, Wientjes CA, Mallant-Hent RC, Siersema PD, Tytgat K, Tuynman H, Kuiken SD, Houben G, Stokkers P, Moons L, Bossuyt P, Fockens P, Mundt MW, Dekker E. Adenoma detection with Endocuff colonoscopy versus conventional colonoscopy: a multicentre randomised controlled trial. Gut. 2017 Mar;66(3):438-445. doi: 10.1136/gutjnl-2015-310097. Epub 2015 Dec 16. PMID 26674360
- [Background] Adler A, Aminalai A, Aschenbeck J, Drossel R, Mayr M, Scheel M, Schroder A, Yenerim T, Wiedenmann B, Gauger U, Roll S, Rosch T. Latest generation, wide-angle, high-definition colonoscopes increase adenoma detection rate. Clin Gastroenterol Hepatol. 2012 Feb;10(2):155-9. doi: 10.1016/j.cgh.2011.10.026. Epub 2011 Nov 2. PMID 22056301
- [Background] Adler A, Aschenbeck J, Yenerim T, Mayr M, Aminalai A, Drossel R, Schroder A, Scheel M, Wiedenmann B, Rosch T. Narrow-band versus white-light high definition television endoscopic imaging for screening colonoscopy: a prospective randomized trial. Gastroenterology. 2009 Feb;136(2):410-6.e1; quiz 715. doi: 10.1053/j.gastro.2008.10.022. Epub 2008 Oct 15. PMID 19014944
- [Background] Adler A, Lieberman D, Aminalai A, Aschenbeck J, Drossel R, Mayr M, Mross M, Scheel M, Schroder A, Keining C, Stange G, Wiedenmann B, Gauger U, Altenhofen L, Rosch T. Data quality of the German screening colonoscopy registry. Endoscopy. 2013 Oct;45(10):813-8. doi: 10.1055/s-0033-1344583. Epub 2013 Sep 9. PMID 24019130
- [Background] Adler A, Pohl H, Papanikolaou IS, Abou-Rebyeh H, Schachschal G, Veltzke-Schlieker W, Khalifa AC, Setka E, Koch M, Wiedenmann B, Rosch T. A prospective randomised study on narrow-band imaging versus conventional colonoscopy for adenoma detection: does narrow-band imaging induce a learning effect? Gut. 2008 Jan;57(1):59-64. doi: 10.1136/gut.2007.123539. Epub 2007 Aug 6. PMID 17681999
- [Background] Adler A, Roll S, Marowski B, Drossel R, Rehs HU, Willich SN, Riese J, Wiedenmann B, Rosch T; Berlin Private-Practice Gastroenterology Working Group. Appropriateness of colonoscopy in the era of colorectal cancer screening: a prospective, multicenter study in a private-practice setting (Berlin Colonoscopy Project 1, BECOP 1). Dis Colon Rectum. 2007 Oct;50(10):1628-38. doi: 10.1007/s10350-007-9029-y. PMID 17694415
- [Background] Adler A, Wegscheider K, Lieberman D, Aminalai A, Aschenbeck J, Drossel R, Mayr M, Mross M, Scheel M, Schroder A, Gerber K, Stange G, Roll S, Gauger U, Wiedenmann B, Altenhofen L, Rosch T. Factors determining the quality of screening colonoscopy: a prospective study on adenoma detection rates, from 12,134 examinations (Berlin colonoscopy project 3, BECOP-3). Gut. 2013 Feb;62(2):236-41. doi: 10.1136/gutjnl-2011-300167. Epub 2012 Mar 22. PMID 22442161
- [Background] Aminalai A, Rosch T, Aschenbeck J, Mayr M, Drossel R, Schroder A, Scheel M, Treytnar D, Gauger U, Stange G, Simon F, Adler A. Live image processing does not increase adenoma detection rate during colonoscopy: a randomized comparison between FICE and conventional imaging (Berlin Colonoscopy Project 5, BECOP-5). Am J Gastroenterol. 2010 Nov;105(11):2383-8. doi: 10.1038/ajg.2010.273. Epub 2010 Jul 13. PMID 20628363
- [Background] Schachschal G, Mayr M, Treszl A, Balzer K, Wegscheider K, Aschenbeck J, Aminalai A, Drossel R, Schroder A, Scheel M, Bothe CH, Bruhn JP, Burmeister W, Stange G, Bahr C, Kiesslich R, Rosch T. Endoscopic versus histological characterisation of polyps during screening colonoscopy. Gut. 2014 Mar;63(3):458-65. doi: 10.1136/gutjnl-2013-304562. Epub 2013 Jun 28. PMID 23812324
- [Background] Schachschal G, Sehner S, Choschzick M, Aust D, Brandl L, Vieth M, Wegscheider K, Baretton GB, Kirchner T, Sauter G, Rosch T. Impact of reassessment of colonic hyperplastic polyps by expert GI pathologists. Int J Colorectal Dis. 2016 Mar;31(3):675-83. doi: 10.1007/s00384-016-2523-8. Epub 2016 Feb 4. PMID 26847619
- [Derived] Zimmermann-Fraedrich K, Sehner S, Rosch T, Aschenbeck J, Schroder A, Schubert S, Liceni T, Aminalai A, Spitz W, Mohler U, Heller F, Berndt R, Bartel-Kowalski C, Niemax K, Burmeister W, Schachschal G. Second-generation distal attachment cuff for adenoma detection in screening colonoscopy: a randomized multicenter study. Gastrointest Endosc. 2023 Jan;97(1):112-120. doi: 10.1016/j.gie.2022.08.030. Epub 2022 Aug 27. PMID 36030888